CLINICAL TRIAL: NCT03745846
Title: A Phase 2 Trial to Evaluate the Efficacy and the Safety of Composite Gel Containing Black Raspberry Extract in Removing HPV From Patients With Cervical Intraepithelial Neoplasia(CIN) After Cervical Conization
Brief Title: A Efficacy and Safety Study of Composite Gel Containing Black Raspberry Extract in Removing HPV From Patients With Cervical Intraepithelial Neoplasia(CIN) After Cervical Conization
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIN-HPV-001
Record Dates: First submitted 2018-11-13; First posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Cervical Intraepithelial Neoplasia; HPV
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Composite Gel Containing Black Raspberry (Experimental): Drug:Composite Gel Containing Black Raspberry 3,000mg Dosage and duration: 1 preparation every other day for 3 months.
  Interventions: Biological: Composite Gel Containing Black Raspberry
- Composite Gel Containing Black Raspberry-placebo (Placebo Comparator): Drug:Composite Gel Containing Black Raspberry-placebo 3,000mg Dosage and duration: 1 preparation every other day for 3 months.
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: Composite Gel Containing Black Raspberry — Composite Gel Containing Black Raspberry 3,000/preparation
  Arms: Composite Gel Containing Black Raspberry
Biological: placebo — Composite Gel Containing Black Raspberry-placebo
  Arms: Composite Gel Containing Black Raspberry-placebo

SUMMARY:
To evaluate the efficacy and safety of composite gel containing black raspberry extract in removing HPV From patients With cervical intraepithelial neoplasia(CIN) after cervical conization

DETAILED DESCRIPTION:
A large number of basic research and animal experiments have confirmed that black raspberry and its active ingredients are used for chemo-prevention of tumors. In recent years, it has been reported that black raspberry extract can effectively inhibit the proliferation of human oral cancer cells and colorectal cancer cells and promote its apoptosis. At the same time, studies have found that chemically modified lactoglobulin exhibits highly potent antiviral activity against human papillomavirus (HPV) infection, including HPV6, HPV16 and HPV18, and can be used as an effective and safe antiviral drug for treatment and Prevent HPV infection. This study attempts to apply black raspberry and lactoglobulin to remove HPV virus and prevent cervical cancer, in order to make breakthroughs in the prevention and control of cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were able and willing to sign informed consent.
* Patients with CIN who underwent cervical conization were at high risk of persistent HPV infection.
* Age must be between 20-55 years old.
* Subjects should begin receiving protocol studies at least two months after cervical conization.
* Patients must be readily available for study and follow-up.
* Patients should not participate in other clinical trials at the same time and agree not to participate in other interventional clinical trials during the protocol study. Except for questionnaires or observational studies.
* Patients should have appropriate nutritional status: body mass index BMI ≥ 18 kg / m2, body weight > 40 kg, serum albumin ≥ 3 g / dL.

Exclusion Criteria:

Anyone who meets any of the following criteria is not allowed to participate in this test:

* Pregnant women, pregnant and lactating women.
* Patients who participated in other clinical trials in the past 3 months.
* It has a serious primary disease such as cardiovascular and cerebrovascular, hematopoietic system and liver and kidney, or patients with mental illness.
* Allergic patients.
* People with epidemics such as AIDS.
* Suffering from uncontrolled complications, including but not limited to: persistent or active infection; clinically significant healing or non-healing wounds; symptomatic congestive heart failure; unstable angina; clinically significant arrhythmia; A disease that affects research compliance, such as an infectious disease or a mental illness/social condition.
* Active, uncontrolled bacterial, viral or fungal infections and require systemic treatment.
* The patient has a history of other malignancies or is suffering from malignant tumors and autoimmune diseases.
* Have any active disease that may increase the risk of a program study or impair a patient's ability to receive protocol research.
* Patients who plan to stay on vacation for 14 days or more during the study period.

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
negative rate | 3 months
  the effective rate and clearance rate of HPV infection from baseline as compared to placebo

SECONDARY OUTCOMES:
Adverse Events | 3 months
  The Rate of Solicited Adverse Events and the Related Features
recurrence rate | 3 months
  The recurrence rate after HPV clearance was assessed